CLINICAL TRIAL: NCT02850302
Title: Triple Negative Breast Cancer: Identification Pilot Study of Predictive Transcriptome Profiles of Early Tumor Drug Resistance Observed in 18F-Fluorodeoxyglucose (FDG) PET
Acronym: TRANSTEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TRANSTEP
Record Dates: First submitted 2016-07-25; First posted 2016-08-01 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FDG PET + exome analysis before treatment and after (Other): Participants will performed one PET with FDG an tumor exome analysis before treatment is started.After 6 cycles of chemotherapy a second PET with FDG and a second tumor exome analysis will be performed
  Interventions: Other: PET with FDG; Other: Tumor exome analysis

INTERVENTIONS:
Other: PET with FDG — A PET with FDG will be performed before the treatment is started and after 6 cycles of chemotherapy.
Other: Tumor exome analysis — A biopsy of the tumor will be performed before the treatment is started and after 6 cycles of chemotherapy. Tumor exome analysis will be performed before treatment is started and after 6 cycles of chemotherapy.

SUMMARY:
Breast cancer is a major public health problem. In France, it is the leading cause of cancer death in women. According to the National Cancer Institute (INCA), approximately 49,000 new cases were diagnosed in 2012 in France.

It is an heterogeneous disease, comprising a plurality of entities whose clinical behavior, biological and prognosis differ. Amongst these entities, the breast cancer triple negative (TN) is defined by the absence of expression of estrogen receptor and progesterone and the absence of overexpression of HER2 oncoprotein. It represents about 15% of breast cancers and occurs more frequently in young women. This is a very proliferative tumor phenotype with metastatic potential. Because of its genomic heterogeneity and lack of recurrent identified molecular target, no targeted therapy has today shown benefit in terms of survival compared to conventional cytotoxic chemotherapy, which partly explains the very poor prognosis of this tumor phenotype. The positron emission tomography (PET) with 18Fluoro-deoxy-glucose (FDG) is a molecular imaging test that can identify from the first or second neoadjuvant chemotherapy treatment non-responder patients to treatment with low probability of pathologic complete response (pCR) after neoadjuvant chemotherapy. For this two FDG-PET examinations should be performed; a) a pretreatment PET b) a control PET after one or two treatments. The objective of this pilot, single-center, prospective study is a preliminary identification of recurrent genomic alterations among triple-negative tumors with early chemoresistance, identified by PET in the first cycle of neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Women more than 18 years old
* breast cancer recently diagnosis (no prior treatment), histologically proven
* stade II or III in the "International union against cancer"(UICC) classification
* non metastatic patient
* Eastern Cooperative Oncology Group (ECOG) 0 or 1
* Negativity of estrogen and progesterone receptor of the tumor (<10%)
* Absence of overexpression of HER2 according to the classification Immunohistochemistry (IHC) - score 0 or 1+
* Patient having read the information note
* written, dated and signed Informed consent

Exclusion Criteria:

* Unresectable breast cancer, bilateral, inflammatory (T4d) or metastatic.
* Unbalanced diabetes during PET scans (glucose more or equal to 9 mmol)
* Small breast cancer indication with first-conserving surgery
* Treated breast cancer history
* Pregnancy or breastfeeding
* Refusal of the patient for trial participation
* Private Person of liberty under supervision or under curators
* Inability to submit to medical follow-up testing for social or psychological reasons
* No affiliation to a social security scheme or medical state aid or the universal medical coverage
* Known allergy or hypersensitivity to 18F-fluorodeoxyglucose
* Patients with known renal impairment (creatinine clearance <60 ml / min / 1.73m2) or a known hepatic failure
* Patients with a strict regime without salt (sodium levels may be higher than 1 mmol in a dose of 18 FDG).

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-11-08 (Actual); Primary Completion 2016-11-08 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Variation of mutational profile | 15 days
  Variation of the mutational profile of the tumor will be assess by exome analysis

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Fumoleau, Pr, Study Director — Centre Georges François Leclerc
Locations (1):
- CGFL, Dijon, France